CLINICAL TRIAL: NCT04381832
Title: A Phase 1b/2, Open-Label, Randomized Platform Study Evaluating the Efficacy and Safety of AB928-Based Treatment Combinations in Patients With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Adenosine Receptor Antagonist Combination Therapy for Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC-6
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-09

CONDITIONS: Prostatic Neoplasms, Castration-Resistant; Androgen-Resistant Prostatic Neoplasms; Castration Resistant Prostatic Neoplasms; Prostatic Cancer, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — zimberelimab; quemliclustat; enzalutamide; Docetaxel; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Stage 1 and 2: Etrumadenant + zimberelimab + enzalutamide (Experimental): Participants will receive oral etrumadenant in combination with intravenous (IV) zimberelimab and standard oral enzalutamide
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab; Drug: Enzalutamide
- Stage 2: enzalutamide (Active Comparator): Participants will receive standard oral enzalutamide
  Interventions: Drug: Enzalutamide
- Stage 1 and 2: Etrumadenant + zimberelimab + docetaxel (Experimental): Participants will receive oral etrumadenant in combination with IV zimberelimab and standard IV docetaxel
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab; Drug: Docetaxel
- Stage 2: docetaxel (Active Comparator): Participants will receive standard dose of IV docetaxel
  Interventions: Drug: Docetaxel
- Stage 1 and 2: Etrumadenant + zimberelimab (Experimental): Oral etrumadenant in combination IV zimberelimab
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab
- Stage 2: Etrumadenant + zimberelimab + quemliclustat (Experimental): Participants will receive oral etrumadenant in combination with IV zimberelimab and IV quemliclustat
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab; Drug: Quemliclustat
- Stage 2: Etrumadenant + quemliclustat (Experimental): Participants will receive oral etrumadenant in combination with IV quemliclustat
  Interventions: Drug: Etrumadenant; Drug: Quemliclustat
- Stage 1: Etrumadenant + zimberelimab PK Sub-Study (Experimental): Participants will receive oral etrumadenant in combination with IV zimberelimab
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab
- Stage 1 and 2: Etrumadenant + SG (Experimental): Participants will receive oral etrumadenant in combination with IV SG.
  Interventions: Drug: Etrumadenant; Drug: SG
- Stage 1 and 2: Etrumadenant + Zimberelimab + SG (Experimental): Participants will receive oral etrumadenant in combination with IV zimberelimab and SG.
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab; Drug: SG

INTERVENTIONS:
Drug: Etrumadenant — Etrumadenant is an A2aR and A2bR antagonist
  Other Names: AB928
  Arms: Stage 1 and 2: Etrumadenant + SG; Stage 1 and 2: Etrumadenant + Zimberelimab + SG; Stage 1 and 2: Etrumadenant + zimberelimab; Stage 1 and 2: Etrumadenant + zimberelimab + docetaxel; Stage 1 and 2: Etrumadenant + zimberelimab + enzalutamide; Stage 1: Etrumadenant + zimberelimab PK Sub-Study; Stage 2: Etrumadenant + quemliclustat; Stage 2: Etrumadenant + zimberelimab + quemliclustat
Drug: Zimberelimab — Zimberelimab is an anti-PD-1 antibody
  Other Names: AB122
  Arms: Stage 1 and 2: Etrumadenant + Zimberelimab + SG; Stage 1 and 2: Etrumadenant + zimberelimab; Stage 1 and 2: Etrumadenant + zimberelimab + docetaxel; Stage 1 and 2: Etrumadenant + zimberelimab + enzalutamide; Stage 1: Etrumadenant + zimberelimab PK Sub-Study; Stage 2: Etrumadenant + zimberelimab + quemliclustat
Drug: Quemliclustat — Quemliclustat is a Cluster of Differentiation (CD)73 Inhibitor.
  Other Names: AB680
  Arms: Stage 2: Etrumadenant + quemliclustat; Stage 2: Etrumadenant + zimberelimab + quemliclustat
Drug: Enzalutamide — Enzalutamide is an androgen receptor inhibitor
  Other Names: Xtandi
  Arms: Stage 1 and 2: Etrumadenant + zimberelimab + enzalutamide; Stage 2: enzalutamide
Drug: Docetaxel — Docetaxel is type of chemotherapy
  Other Names: Taxotere
  Arms: Stage 1 and 2: Etrumadenant + zimberelimab + docetaxel; Stage 2: docetaxel
Drug: SG — Sacituzumab govitecan is an antibody-drug conjugate
  Other Names: Trodelvy
  Arms: Stage 1 and 2: Etrumadenant + SG; Stage 1 and 2: Etrumadenant + Zimberelimab + SG

SUMMARY:
This is a Phase 1b/2, open-label, multicenter platform trial to evaluate the antitumor activity and safety of etrumadenant (AB928)-based combination therapy in participants with metastatic castrate resistant prostate cancer (mCRPC).

ELIGIBILITY:
General Inclusion Criteria:

* Male participants; age ≥ 18 years
* Metastatic castrate-resistant prostate cancer while on anti-androgen treatment with castrate levels of testosterone (≤1.7 nanomoles per liter [nmol/L] or 50 nanograms per deciliter [ng/dL])
* Measurable or non-measurable disease as per radiographic evaluation
* Participants with measurable disease may require a fresh tumor biopsy at study entry
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Life expectancy of at least 3 months
* Adequate hematologic and end-organ function
* Human immunodeficiency virus (HIV), Hepatitis B, and C test results negative prior to first study treatment

Inclusion Criteria for Participants receiving an enzalutamide-containing treatment

* Disease progression after prior treatment with abiraterone

Inclusion Criteria for Participants receiving a docetaxel-containing treatment

* Disease progression after prior androgen synthesis inhibitor therapy

Inclusion Criteria for all other Participants

* Disease progression after prior androgen synthesis inhibitor treatment and up to 2 prior lines of taxane chemotherapy

General Exclusion Criteria:

* Prior treatment with immune checkpoint blockade therapy
* Prior anticancer treatment including approved agents, systemic radiotherapy, or investigational therapy, within 2-4 weeks prior first study treatment
* Corrected QT interval (QTc) ≥480 msec using Fredericia's QT correction formula (based on an average of triplicate recordings)
* Prior allogeneic stem cell or solid organ transplantation
* Prior treatment with drugs that stimulate the immune system within 4 weeks prior to first study treatment
* Prior treatment with drugs that suppress the immune system within 2 weeks prior to first study treatment
* Received a live, attenuated vaccine within 4 weeks prior to first study treatment, or may need to receive a vaccine during study treatment
* Presence of metastases in the brain or cancer spreading into the cerebrospinal fluid - CSF (leptomeningeal disease)
* Prior pulmonary fibrosis, pneumonia, or pneumonitis
* Cancer other than prostate within 2 years prior to study entry, except for some cancers with a low risk of spreading like non-melanoma skin
* Prior treatment with an agent targeting the adenosine pathway
* No oral or IV antibiotics within 2 weeks prior to first study treatment
* No severe infection within 4 weeks prior to first study treatment
* No clinically significant cardiac disease
* Inability to swallow medications

Exclusion Criteria for Participants receiving an enzalutamide-containing treatment

* Prior treatment with docetaxel, cabazitaxel, or other taxane chemotherapy (prior docetaxel [up to 6 cycles] for hormone-sensitive prostate cancer is allowed if the last dose was at least 6 months prior to study treatment initiation)
* Prior treatment with enzalutamide or similar therapy other than abiraterone
* Active or history of autoimmune disease or immune deficiency
* History of severe allergic reactions to antibody therapy
* Concomitant use of a medication prohibited by the protocol (including certain transporter substrates as well as known strong CYP3A4 inducers and CYP3A4 inhibitors) within 4 weeks prior to and throughout study treatment

Exclusion Criteria for Participants receiving a docetaxel-containing treatment

* Prior treatment with docetaxel, cabazitaxel, or other taxane chemotherapy
* Active or history of autoimmune disease or immune deficiency
* History of severe allergic reactions to antibody therapy
* Concomitant use of a medication prohibited by the protocol (including certain transporter substrates as well as known strong CYP3A4 inducers and CYP3A4 inhibitors) within 4 weeks prior to and throughout study treatment

Exclusion Criteria for all other Participants

* Prior treatment with docetaxel, cabazitaxel, topoisomerase 1 inhibitors, or other taxane chemotherapy
* Active or history of autoimmune disease or immune deficiency
* History of severe allergic reactions to antibody therapy
* Concomitant use of a medication prohibited by the protocol (including certain transporter substrates as well as known strong CYP3A4 inducers and CYP3A4 inhibitors) within 4 weeks prior to and throughout study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in Stage 1 and 2 | From study enrolment until participant discontinuation, or first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 3-5 years)
  ORR defined as the composite proportion of participants with a Prostate Specific Antigen (PSA) and/or radiographic complete response (CR) and partial response (PR) determined by the investigator according to the Prostate Cancer Working Group 3 (PCWG3) criteria
Incidence and Severity of AEs and Serious Adverse Events (SAEs) in Stage 1 | From first dose date to 90 days after the last dose (approximately 1.5 years)

SECONDARY OUTCOMES:
Percentage of participants with a PSA response in Stage 1 and 2 | From study enrollment until disease progression or loss of clinical benefit (approximately 3-5 years)
  PSA response defined as the proportion of participants with a confirmed PSA decrease from baseline of 50% or more based on two consecutive assessments measured 3 to 4 weeks apart
Percentage of participants with Radiographic Response in Stage 1 and 2 | From study enrollment until disease progression or loss of clinical benefit (approximately 3-5 years)
  Radiographic Response is measurable disease at baseline who achieved a best overall response of CR or PR according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Percentage of Participants with Disease Control Rate in Stage 1 and 2 | From study enrollment until disease progression or loss of clinical benefit (approximately 3-5 years)
  Disease Control Rate is defined as the percentage of participants with measurable disease at baseline who achieved a best overall RECIST response of CR, PR, or Stable Disease (SD).
Serum/Plasma Concentration for etrumadenant, zimberelimab, and enzalutamide when administered as part of a combination regimen in Stage 1 and 2. | Recorded at baseline (enrollment), during the first 5 months of treatment and 3 additional timepoints in the first year of treatment. (approximately 1.5 years)
Serum/Plasma Concentration for etrumadenant and zimberelimab when administered as part of a combination regimen with docetaxel in Stage 1 and 2 | Recorded at baseline (enrollment), during the first 5 months of treatment and 3 additional timepoints in the first year of treatment. (approximately 1.5 years)
Serum/Plasma Concentration for etrumadenant and zimberelimab when administered as part of a combination regimen in Stage 1 and 2 | Recorded at baseline (enrollment), during the first 5 months of treatment and 3 additional timepoints in the first year of treatment. (approximately 1.5 years)
Serum/Plasma Concentration for etrumadenant, zimberelimab, and AB680 when administered as part of a combination regimen in Stage 1 and 2 | Recorded at baseline (enrollment), during the first 5 months of treatment and 3 additional timepoints in the first year of treatment. (approximately 1.5 years)
Serum/Plasma Concentration for etrumadenant and AB680 when administered as part of a combination regimen in Stage 1 and 2. | Recorded at baseline (enrollment), during the first 5 months of treatment and 3 additional timepoints in the first year of treatment. (approximately 1.5 years)
Percentage of participants with anti-drug antibodies to zimberelimab in Stage 1 and 2 | Recorded at baseline (enrollment), during the first 4 months of treatment, 4 additional timepoints in the first year of treatment, and at end of treatment. (approximately 1.5 years)
Incidence and severity of AEs and serious adverse events (SAEs) in Stage 2 | From first dose date to 90 days after the last dose (approximately 3-5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (19):
- United States (17):
  - The Oncology Institute of Hope & Innovation, Cerritos, California
  - The University of California, Los Angeles, Encino, California
  - The University of California, Irvine Medical Center, Orange, California
  - Florida Cancer Specialists South, Sarasota, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Florida Cancer Specialists Panhandle, Tallahassee, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Affinity Health Hope & Healing Cancer Services, Hinsdale, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - New York University, Langone Health, New York, New York
  - Wilmot Cancer Institute Oncology, University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Medical Oncology Associates, PS (dba Summit Cancer Centers), Spokane, Washington
- Canada (2):
  - Juravinski Cancer Center, Hamilton, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM) Centre de Recherche, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy